CLINICAL TRIAL: NCT00126035
Title: Open, Randomised, Multi-Centre, Cross-Over Study to Investigate the Efficacy of the Migraid Device Compared With No Device Treatment in the Acute, Early Treatment of Migraine With Typical Aura
Brief Title: Study With Migraid Device in Acute, Early Treatment of Migraine With Typical Aura
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Profess Medical Consultancy (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 03-MIG-01
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 2005-07

CONDITIONS: Migraine With Typical Aura
Keywords: Acute Migraine; Device; Migraid; Treatment; Aura
MeSH Terms: conditions — Migraine with Aura; Epilepsy

INTERVENTIONS:
Device: Migraid

SUMMARY:
The purpose of the study was to assess the efficacy of Migraid in terms of preventing headaches in patients with migraine with typical aura. The secondary objectives were to assess whether Migraid is able to achieve pain relief and/or relief of migraine associated symptoms and to evaluate the safety and tolerability of the study treatment.

DETAILED DESCRIPTION:
Migraid is to be used only once during the aura phase of a migraine attack for a duration of 60 minutes.

Reference therapy: No treatment. This means that at random the patient will be allocated to either of the two treatment orders; the first treatment order is to use the Migraid whenever a migraine attack with an aura occurs. During the next migraine attack the Migraid will not be used and vice versa for the other group of patients.

Patients will be asked to complete diary cards to record details for each of the two migraine attacks and the severity of the migraine headache at certain points in time: at t = 30 minutes, t = 60 minutes, t= 90 minutes, t =120 minutes, t =150 minutes, t =180 minutes and t = 24 hours.

Also, associated symptoms will be asked for. Rescue medication data including name, time taken and amount will also be registered in the diary card.

For all primary and secondary variables of efficacy, the following definitions will be used:

Grade or score: Pain level: Description

0: None - No pain;

1. Mild - A headache with no remarkable pain that does not hinder you in performing your usual daily activities;
2. Moderate - A headache with pain that hinders you in performing your usual daily activities, but that does necessitate you to go to bed;
3. Severe - A headache with pain that necessitates you to go to or stay in bed.

The associated symptoms will be graded as either present or absent. These symptoms are defined to conform to the following table:

Symptom: Description

Nausea: Sick to the stomach/feel like throwing up; Vomiting: Throwing up or puking; Photophobia: Light bothers or hurts the eyes; Phonophobia: Noise bothers or hurts the ears.

A migraine attack is defined as:

New onset of migraine pain, preceded by a pain-free period of at least 24-hours duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a current history of migraine with typical aura where the aura is usually followed by headache according to the International Headache Society (IHS) criteria.
* Patients are male or female. N.B. When female patients are treated for migraine attacks with triptans then the required precautions and safety measures should be taken in order to prevent pregnancy.
* Patients with an age between 18 and 65 years.
* Patients must have experienced 1-4 moderate (grade 2) or severe (grade 3) migraine attacks per month for at least two months prior to entry into the study.
* Patients must be willing to keep their prophylactic drug treatment for migraine unchanged.
* Patients must be able to distinguish migraine headaches from other headache types (e.g. tension-type headaches) at the onset of a migraine attack.
* Patients must be able to understand and complete the diary card
* Patients must be willing and able to give written informed consent prior to entry into the study.
* Patients must be willing and able to carry the Migraid and, if necessary, apply it in a public place.

Exclusion Criteria:

* Migraine patients with a typical aura but without any migraine headache thereafter.
* Patients with a history suggestive of ischaemic heart disease (IHD) or any present evidence of ischaemic heart disease (like angina pectoris, previous myocardial infarction, documented silent ischaemia, Prinzmetal's angina), or symptoms consistent with IHD.
* Patients suffering from coronary vasospasm or any atherosclerotic disease (cerebrovascular disease [CVD], peripheral vascular disease [PVD] or Raynaud's disease) which places them at increased risk of coronary ischaemia.
* Patients with a history of cerebrovascular accident (CVA) or transient ischaemic attacks (TIA).
* Patients with a supine diastolic blood pressure of > 95 mm Hg and/or systolic blood pressure > 160 mm Hg (treated or untreated) at Visit 1.
* Patients with a history of epilepsy or structural brain lesions which lower their convulsion threshold.
* Patients with tension-type headaches > 15 days/month in either of the two months prior to the study.
* Current abuse of opioid analgesics or other psychotropic drugs. History (within the past year) or current abuse of ergotamine (abuse as defined as > 10 mg/week). Current abuse of alcohol (according to local recommendations) or other drugs.
* Patients suffering from any severe concurrent medical condition which may affect the interpretation of efficacy and safety data or which otherwise contraindicates participation in a clinical study.
* Patients with a history of ophthalmoplegic, basilar or hemiplegic migraine.
* Patients with a history of impaired hepatic or renal function.
* Patients who have participated in a clinical trial within the previous 3 months or are planning to participate in another clinical research study at any time during this study.
* Patients with any concurrent medical or psychiatric condition that, in the investigator's opinion, may affect the interpretation of efficacy or safety data or which otherwise contraindicates participation in a clinical trial.
* Patients cannot be participating investigators, study co-ordinators, employees of investigators, or family members of any of the aforementioned.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134
Dates: Start 2004-02; Study Completion 2004-12

PRIMARY OUTCOMES:
Percentage of attacks that were "pain free" at t = 120 minutes without using rescue medication

SECONDARY OUTCOMES:
Percentage of responders
Percentage of attacks that were "pain free" at t = 30 minutes, t = 60 minutes, t = 90 minutes, t =150 minutes, t =180 minutes and t = 24 hours without using rescue medication
Percentage of attacks that were "sustained pain free" without using rescue medication
Percentage of attacks resulting in "headache relief" at t = 60 minutes, t = 90 minutes, t =120 minutes, t =150 minutes, t =180 minutes and t = 24 hours without using rescue medication
Percentage of attacks resulting in "sustained headache relief" without using rescue medication
Percentage of attacks with relief of nausea and vomiting, photo- and phonophobia at t = 30 minutes, t = 60 minutes, t = 90 minutes, t = 120 minutes, t=180 minutes and t = 24 hours without using rescue medication
Percentage of attacks with return of headache without using rescue medication
Percentage of attacks for which the patient's usual rescue medication is taken
Patient preference, as well as reasons for preference

CONTACTS AND LOCATIONS:
Overall Officials: Joop AM Kuster, MD, Principal Investigator — Kennemer Gasthuis Hospital
Locations (1):
- Multicentre study with 21 General practitioners, Haarlem, North Holland, Netherlands

REFERENCES:
- See also: new website for the Migraid device — http://www.migraid.com